CLINICAL TRIAL: NCT05026905
Title: A Phase II Randomized Study of Gemcitabine and Nab-paclitaxel in Combination With S- 1/LV (GASL) or Oxaliplatin (GAP) as First-line Treatment for Metastatic Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: T5221
Record Dates: First submitted 2021-08-24; First posted 2021-08-30 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Phase II, Open-label, Parallel 2-arm, Multi-center
Keywords: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; 130-nm albumin-bound paclitaxel; S 1 (combination); Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GASL arm (Other): eligible patients will receive gemcitabine 800 mg/m2 on day 1, nab-paclitaxel 125 mg/m2 on day 1, S-1 orally 60-100 mg/day [depending on patient's baseline body surface area (BSA)] on day 1 to 7 and leucovorin 30mg BID day 1 to 7 on in a 2-week cycle. The dose of S-1 is defined as follows:
  * BSA < 1.25 m2: 60 mg/day
  * 1.25 m2 ≤ BSA < 1.5 m2: 80 mg/day
  * BSA ≥ 1.5 m2: 100 mg/day
  Interventions: Drug: Gemcitabine 1000 mg; Drug: Nab paclitaxel; Drug: S1; Drug: leucovorin
- GAP arm (Other): eligible patients will receive gemcitabine 800 mg/m2, nab-paclitaxel 125 mg/m2 and oxaliplatin 75mg/m2 on day 1 in a 2-week cycle.
  Interventions: Drug: Gemcitabine 1000 mg; Drug: Nab paclitaxel; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine 1000 mg — Gemcitabine 800mg/m2 in N/S 250ml over 30 minutes (or fixed dose rate 10 mg/m2/min) IV infusion on day 1 repeated every 14 days.
  Other Names: Gemcitabine
Drug: Nab paclitaxel — Nab-paclitaxel 125mg/m2 over 30 minutes IV infusion on day 1 repeated every 14 days, followed by Gemcitabine
  Other Names: nab-paclitaxel
Drug: S1 — S-1 orally 60-100 mg/day day 1 to 7 on in a 2-week cycle. The dose of S-1 is defined as follows:
  * BSA < 1.25 m2: 60 mg/day
  * 1.25 m2 ≤ BSA < 1.5 m2: 80 mg/day
  * BSA ≥ 1.5 m2: 100 mg/day
  Other Names: S-1
  Arms: GASL arm
Drug: leucovorin — leucovorin 30mg BID day 1 to 7 on in a 2-week cycle
  Other Names: Calcium Folinate tablet
  Arms: GASL arm
Drug: Oxaliplatin — Oxaliplatin 75mg/m2 in 250 mL of D5W over 120 minutes IV infusion on day 1 repeated every 14 days
  Arms: GAP arm

SUMMARY:
Gemcitabine and nab-paclitaxel are one standard of care for metastatic pancreatic adenocarcinoma (mPDAC) but the progression free survival (PFS) of the regimen is only 5.5 months. Previous phase II study showed gemcitabine and nab-paclitaxel plus cisplatin had a PFS of 10.1 months in mPDAC. This study will evaluate the efficacy and safety of gemcitabine, nab-paclitaxel plus S-1/LV (GASL) against gemcitabine, nab-paclitaxel plus oxaliplatin (GAP) in patients with mPDAC.

DETAILED DESCRIPTION:
Gemcitabine and nab-paclitaxel are one standard of care for metastatic pancreatic adenocarcinoma (mPDAC) but the progression free survival (PFS) of the regimen is only 5.5 months. Previous phase II study showed gemcitabine and nab-paclitaxel plus cisplatin had a PFS of 10.1 months in mPDAC. However, the nephrotoxicity of cisplatin is always a concern therefore cisplatin was substituted with oxaliplatin in current study. S-1 monotherapy has shown promising anti-tumor activity against PDAC with a manageable safety profile which provided the opportunity of combination with other agents. In this study, we will evaluate the efficacy and safety of gemcitabine, nab-paclitaxel plus S-1/LV (GASL) against gemcitabine, nab-paclitaxel plus oxaliplatin (GAP) in patients with mPDAC.

ELIGIBILITY:
Inclusion Criteria:

* A.Cytology or histology confirmed pancreatic adenocarcinoma with evidence of distant metastasis.Mixed component of other cell type (eg, adenosquamous, adenocarcinoma with neuroendocrine differentiation) is eligible but should notify PI before registration.
* B.No history of prior chemotherapy for pancreatic cancer, except adjuvant chemotherapy that completed at least 6 months before documentation of recurrence by imaging study.
* C.Patients with prior radiotherapy are eligible if there are other measurable target lesions that is not irradiated.
* D.At least one measurable lesion according to RECIST version 1.1
* E.Ability to understand and willingness to sign a written informed consent document.
* F.ECOG performance status 0-1
* G.Age of 20 years or above
* H.Adequate organ function as defined by the following criteria:

absolute neutrophil count (ANC) ≥ 1,500/mm3 hemoglobin level ≥ 9 g/dL platelet count ≥ 100,000/mm3 total bilirubin ≤ 2 ULN or ≤5 ULN if caused by biliary obstruction and achieving adequate drainage judged by investigator aspartate aminotransferase (AST) / alanine aminotransferase (ALT) ≤ 3 x ULN or ≤ 5.0×ULN in the presence of liver metastases creatinine clearance rate (CCr) ≥ 50 mL/min (24-hour urine collection or calculated by Cockroft-Gault formula; male: [(140 - age) × weight (kg)]/[72 × serum creatinine(mg/dL)];female=male x 0.85

-I.Patients with childbearing potential shall have effective contraception for both the patient and his or her partner during the study.

Exclusion Criteria:

* A. Other malignancy within the past 5 years except for adequately treated localized cancer or carcinoma in situ;All patients with other malignancy within the past 5 years should notify PI before registration.
* B.Active or uncontrolled infection;
* C.Significant medical conditions that is contraindicated to study medication or render patient at high risk from treatment complications at physician discretion
* D.Pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential.
* E.History of active autoimmune disease within 3 years or use of steroid more than prednisolone 10mg/day.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-12-28 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Best objective response rate (ORR) | 6 years
  tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 6 years
  Defined as having complete response, partial response or stable disease at least 12 weeks.
Progression-free survival (PFS) | 6 years
  from the start date of study treatment to the date of progression disease or death.
Overall survival (OS) | 6 years
  from the start date of study treatment to the date of death.
Duration of response (DOR) | 6 years
  time from documentation of tumor response to disease progression.
Incidence of Treatment-related Adverse Events [Safety and Tolerability] | 6 years
  This study will utilize the NCI-CTCAE v5.0 for Adverse Event monitoring and reporting

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD, Ph.D., Study Chair — National Health Research Institutes, Taiwan; Yung-Yeh Su, M.D., Principal Investigator — National Health Research Institutes, Taiwan; Shang-Hung Chen, M.D., Principal Investigator — National Health Research Institutes, Taiwan
Locations (4):
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No